CLINICAL TRIAL: NCT01477320
Title: Enteral Nutrition as Stress Ulcer Prophylaxis in Critically Ill Patients. Prospective, Double-blind, Randomized, Placebo-controlled Study.
Brief Title: Enteral Nutrition as Stress Ulcer Prophylaxis in Critically Ill Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed Saad (Other)
Collaborators: Abbott Nutrition (Industry); University of Louisville (Other)
Responsible Party: Sponsor-Investigator, Mohamed Saad, Primary Investigator, University of Louisville
Organization: University of Louisville (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 11.0170
Record Dates: First submitted 2011-10-04; First posted 2011-11-22 (Estimated); Results first posted 2018-01-16 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2017-12

CONDITIONS: Gastrointestinal Hemorrhage; Clostridium Difficile Colitis
Keywords: Enteral Nutrition; Stress Ulcer Prophylaxis; Critically Ill Patients; Overt and significant GI bleeding; Stress gastropathy; Clostridium Difficile pseudomembranous colitis; Vital AF; Small peptide fish oil structured lipids; Fructose oligosaccharide
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Enterocolitis, Pseudomembranous | interventions — Pantoprazole; Enteral Nutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pantoprazole 40mg IV daily and tube feed (Active Comparator)
  Interventions: Drug: Pantoprazole 40 mg IV daily and tube feed.
- Placebo and tube feed. (Placebo Comparator)
  Interventions: Other: Placebo and tube feed

INTERVENTIONS:
Drug: Pantoprazole 40 mg IV daily and tube feed. — Patients randomized to the control group "active Comparator" will receive tube feed plus an Pantoprazole 40 mg IV daily.
  Other Names: Tube feed formula:(Vital AF "Advanced Formula" 1.2 Cal(TM),Abbott,Columbus,OH)
  Arms: Pantoprazole 40mg IV daily and tube feed
Other: Placebo and tube feed — Patients randomized to Placebo group "placebo Comparator" will receive tube feed plus an Placebo.
  Other Names: Tube feed formula:(Vital AF "Advanced Formula" 1.2 Cal(TM),Abbott,Columbus,OH)
  Arms: Placebo and tube feed.

SUMMARY:
study is to determine if proton pump inhibitors plus enteral nutrition is superior to enteral nutrition alone as a stress ulcer prophylaxis strategy in critically ill patients in terms of incidence of overt and significant GI bleeding related to stress gastropathy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Admission to the medical ICU at University of Louisville Hospital or Jewish Hospital
* Expected need for mechanical ventilation > 48 hours
* No contraindication to EN within the first 24 hours after admission to the ICU

Exclusion Criteria:

* Evidence of active GI bleeding during current hospitalization prior to study entry
* Admission to ICU with primary diagnosis of burn injury
* Closed head injury or increased intracranial pressure
* Partial or complete gastrectomy
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2013-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Saad, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville hospital, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started in July 2013 in the medical ICU of University of Louisville Hospital. In July 2014, a second recruitment site (medical ICU at Jewish Hospital) was added as a second site for recruitment.
Period: Overall Study
Arm/Group | Pantoprazole 40mg IV Daily and Tube Feed | Placebo and Tube Feed.
Started | 62 | 62
Completed | 55 | 47
Not Completed | 7 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pantoprazole 40mg IV Daily and Tube Feed | Placebo and Tube Feed. | Total
Number analyzed (Participants) | 55 | 47 | 102
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: The patient excluded from analysis were extubated too soon after enrollment before starting tube feed
  years | 62 [49.5 to 68] | 58 [40.5 to 66.5] | 60 [40.5 to 68.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 19 | 44
  Male | 30 | 28 | 58
Region of Enrollment [Number; unit: participants]
  United States | 55 | 47 | 102

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With GI Bleeding
Description: 1. Incidence of overt GI bleeding (as defined by the presence of coffee ground emesis, hematemesis of bright red blood, melena, or hematochezia) seen with Proton Pump Inhibitor (PPI) and EN versus EN alone in critically ill patients.
  2. Incidence of significant GI bleeding, defined by a 3-point decrease in hematocrit within 24 hours accompanied by signs of overt GI bleeding, or by an unexplained 6-point decrease in hematocrit during any 48 hour period.
Time Frame: Subjects will be followed from date of randomization until discharge from the ICU or cessation of Enteral Nutrition (EN) and successful initiation of oral feeds up to 100 weeks.
Measure: Number; unit: participants
Arm/Group | Pantoprazole 40mg IV Daily and Tube Feed | Placebo and Tube Feed.
Number analyzed (Participants) | 55 | 47
participants | 1 | 1

2. Secondary Outcome: Number of Subjects With ICU-acquired C. Difficile Pseudomembranous Colitis.
Time Frame: Subjects will be followed until discharge from the ICU or cessation of EN and successful initiation of oral feeds up to 100 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Pantoprazole 40mg IV Daily and Tube Feed | Placebo and Tube Feed.
Number analyzed (Participants) | 55 | 47
Participants | 1 | 3

ADVERSE EVENTS:
Arm/Group | Pantoprazole 40mg IV Daily and Tube Feed | Placebo and Tube Feed.
Serious Adverse Events (participants affected / at risk) | 1/62 | 1/62
Other Adverse Events (participants affected / at risk) | 0/62 | 0/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pantoprazole 40mg IV Daily and Tube Feed (N=62) | Placebo and Tube Feed. (N=62)
GI bleed (Gastrointestinal disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No